CLINICAL TRIAL: NCT02427503
Title: Sinonasal Functional Impact of Endoscopic Surgery for Bilateral Polyposis on Bronchial Inflammation, Control and Lung Function in Asthma
Brief Title: ATP Project (Asthma afTer Polypectomy)
Acronym: ATP
Status: Completed | Type: Observational
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Universitat Autonoma de Barcelona (Other); Sociedad Española de Neumología y Cirugía Torácica (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-PEN-2015-11
Record Dates: First submitted 2015-03-25; First posted 2015-04-28 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Asthma; Nasal Polyps
Keywords: asthma; sinonasal polyposis; eosinophilic bronchial inflammation; endoscopic sinus surgery
MeSH Terms: conditions — Asthma; Nasal Polyps

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Asthma with NP and require surgery: Patients receiving standardized treatment for nasal polyposis, according to the POLINA guidelines and for persistent asthma who will undergo FESS-BP.
  Interventions: Procedure: Asthma with NP and require surgery
- Asthma with NP and NOT require surgery: Patients receiving standardized treatment for nasal polyposis, according to the POLINA guidelines and for persistent asthma who will NOT undergo FESS-BP.

INTERVENTIONS:
Procedure: Asthma with NP and require surgery — To evaluate the effect on asthma of functional endoscopic sinus surgery of bilateral sinonasal polyposis in patients diagnosed with persistent asthma and grade II or III sinonasal polyposis.
  Groups: Asthma with NP and require surgery

SUMMARY:
Inflammation of the nasal and bronchial mucosa characterizing rhinitis and asthma are probably manifestations of the same disease. Multiple functional observations, pathogenic and clinical support that assertion. It is noteworthy that most asthma patients, who underwent a nasal endoscopic polypectomy, improve your asthma after surgery. This improvement would be related to the administration of oral steroids that these patients usually receive after surgery, or the disappearance of nasal discomfort caused by nasal polyps to improve ventilation. But this does not explain why this improvement, in some cases lasting for months after the operation, and without receiving oral steroids. It is speculated that severe nasal inflammation due to nasal polyps stimulate the bone marrow to produce more eosinophils, an increased supply of blood eosinophils, and consequently, a major bronchial eosinophilic inflammation, aggravating asthma. However, it is noteworthy that studies have evaluated the clinical impact in asthma after endoscopic nasal polypectomy, are scarce or performed on a small number of cases, the results are inconsistent and do not allow categorically whether or not such positive association. And more importantly, none of them included measurements of airway inflammation and hypothesized relationship between bronchial eosinophilic inflammation and nasal polyposis, aclarar.La remains finding that provides nasal endoscopic polypectomy objective improvement of severe asthma it could be a future therapeutic option to consider in patients with asthma and rhinosinusal polyposis.

DETAILED DESCRIPTION:
Sinonasal polyposis (SP) is a chronic inflammatory disease of the lining of the nasal passages and sinuses, with a prevalence of approximately 2-3% of the general population. The prevalence of asthma in patients diagnosed with SP is much greater than that of the general population and can reach half of the cases and indicate a more severe phenotype and worse control in asthmatic patients without SP. It is possible that the pathophysiologic mechanisms underlying the development of SP and concomitant asthma are the same and both processes can be considered the same disease.

Recommendations of major clinical practice guidelines for the treatment of SP include administration of intranasal topical steroids at high doses, and in subjects who do not respond to this treatment or are more severe, administering a course of systemic steroids orally for 10-14 days or surgical intervention including polypectomy and removal of the diseased mucosa endoscopically, known as functional endoscopic sinus surgery (FESS).

In this context, it is noteworthy that most asthma patients, who underwent functional endoscopic sinus surgery for bilateral polyposis (FESS-BP) stated it dramatically improved their asthma after surgery. This improvement could be related to the effect of oral steroids these patients often receive after surgery, or the disappearance of nasal discomfort caused by nasal polyps as ventilation improves after the intervention. However, these reasons do not sufficiently explain the fact that this improvement, in some cases extends for months after surgery, when patients are no longer receiving oral steroids.

It has been speculated that severe nasal inflammation which involves the presence of nasal polyps would constantly stimulate the bone marrow, causing on the one hand increased production of eosinophils and the other an increase in adhesiveness, and thus, an important eosinophilic bronchial inflammation. This is in line with a usual clinical observation according to which patients with asthma and sinonasal polyposis, often suffer more severe asthma; and severe sinus inflammation is one of the aggravating factors recognized in severe uncontrolled asthma.

However, studies that have assessed the clinical impact in asthma after FESS-BP, are only a few or have been performed on a small number of cases. Consequently, the results are inconsistent and do not allow to categorically establish whether this positive association exists or not. Most importantly, however, none of them included measurements of bronchial inflammation in the study variables, so that the hypothesis of the possible relationship between eosinophilic bronchial inflammation and nasal polyposis remains without having been tested.

Moreover, the finding that the FESS-BP provides an objective improvement of asthma, could be a future therapeutic option to consider in patients with severe asthma and sinonasal polyposis.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes aged ≥ 18 and younger than 70 years diagnosed with persistent asthma (according to GEMA4.0 criteria) (18) and grade II and III bilateral sinonasal polyposis of Lildholdlt (9,19), which, as indicated in routine clinical practice established by an otolaryngologist, will undergo FESS.

Exclusion Criteria:

* Intermittent asthma;
* exacerbation of asthma that required treatment with parenteral steroids one month prior to visit 1;
* concomitance of other chronic respiratory diseases (bronchiectasis, fibrosis, etc.);
* other disabling severe comorbidities in the opinion of the investigators;
* previous noninflammatory sinonasal pathology;
* corticosteroid-dependent patients or managed with other immunomodulatory treatments.
* Patients with a history of previous nasal surgery.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with persistent asthma and grade II and III bilateral sinonasal polyposisand, by voluntary decision of the otolaryngologist and the patient, who will offer alternatives treatment to the candidate patient, following the recommendations of clinical practice guidelines.
  If the patient is indicated in routine clinical practice FESS-BP, will be offer to enter to the study.
  If the patient is NOT indicated in routine clinical practice FESS-BP or reject intervention, will be also offer to enter to the study.
Sampling Method: Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2016-07; Primary Completion 2018-12 (Actual); Study Completion 2019-12-16 (Actual)

PRIMARY OUTCOMES:
Breath inflammation measured by the fractional exhaled nitric oxide (FeNO) | 12 months
  part per billion
Asthma control bases on the ACT Questionnaire (Asthma Control Test) | 12 month
  5-25 points, on 5 is bad control and 25 is the maximun asthma control
Spirometry measure FEV1 | 12 month
  percentage
Sputum and blood test | 12 month
  eosinophils percentage

SECONDARY OUTCOMES:
Nasal, inhalated or oral steroid treatment | 12 months
  micrograms/day
Mini questionnaire of quality of life (MiniAQLQ) | 12 months
  1-7 points
Questionnaire of chonic rhinosinusitis (SNOT 22) | 12 month
  0-5 points

CONTACTS AND LOCATIONS:
Overall Officials: Lorena Soto-Retes, physician, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Lorena Soto-Retes, Barcelona, Spain

REFERENCES:
- [Result] Johansson L, Akerlund A, Holmberg K, Melen I, Bende M. Prevalence of nasal polyps in adults: the Skovde population-based study. Ann Otol Rhinol Laryngol. 2003 Jul;112(7):625-9. doi: 10.1177/000348940311200709. PMID 12903683
- [Result] Klossek JM, Neukirch F, Pribil C, Jankowski R, Serrano E, Chanal I, El Hasnaoui A. Prevalence of nasal polyposis in France: a cross-sectional, case-control study. Allergy. 2005 Feb;60(2):233-7. doi: 10.1111/j.1398-9995.2005.00688.x. PMID 15647046
- [Result] Perez De Llano LA, Gonzalez FC, Anon OC, Perea MP, Caruncho MV, Villar AB; Proyecto Camaron (Control del Asma Mediante el Analisis Regular del Oxido Nitrico). [Relationship between comorbidity and asthma control]. Arch Bronconeumol. 2010 Oct;46(10):508-13. doi: 10.1016/j.arbres.2010.05.008. Epub 2010 Jul 17. Spanish. PMID 20638762
- [Result] Grossman J. One airway, one disease. Chest. 1997 Feb;111(2 Suppl):11S-16S. doi: 10.1378/chest.111.2_supplement.11s. PMID 9042022
- [Result] Braunstahl GJ, Overbeek SE, Kleinjan A, Prins JB, Hoogsteden HC, Fokkens WJ. Nasal allergen provocation induces adhesion molecule expression and tissue eosinophilia in upper and lower airways. J Allergy Clin Immunol. 2001 Mar;107(3):469-76. doi: 10.1067/mai.2001.113046. PMID 11240947
- [Result] Togias A. Rhinitis and asthma: evidence for respiratory system integration. J Allergy Clin Immunol. 2003 Jun;111(6):1171-83; quiz 1184. doi: 10.1067/mai.2003.1592. PMID 12789212
- [Result] Bousquet J, Khaltaev N, Cruz AA, Denburg J, Fokkens WJ, Togias A, Zuberbier T, Baena-Cagnani CE, Canonica GW, van Weel C, Agache I, Ait-Khaled N, Bachert C, Blaiss MS, Bonini S, Boulet LP, Bousquet PJ, Camargos P, Carlsen KH, Chen Y, Custovic A, Dahl R, Demoly P, Douagui H, Durham SR, van Wijk RG, Kalayci O, Kaliner MA, Kim YY, Kowalski ML, Kuna P, Le LT, Lemiere C, Li J, Lockey RF, Mavale-Manuel S, Meltzer EO, Mohammad Y, Mullol J, Naclerio R, O'Hehir RE, Ohta K, Ouedraogo S, Palkonen S, Papadopoulos N, Passalacqua G, Pawankar R, Popov TA, Rabe KF, Rosado-Pinto J, Scadding GK, Simons FE, Toskala E, Valovirta E, van Cauwenberge P, Wang DY, Wickman M, Yawn BP, Yorgancioglu A, Yusuf OM, Zar H, Annesi-Maesano I, Bateman ED, Ben Kheder A, Boakye DA, Bouchard J, Burney P, Busse WW, Chan-Yeung M, Chavannes NH, Chuchalin A, Dolen WK, Emuzyte R, Grouse L, Humbert M, Jackson C, Johnston SL, Keith PK, Kemp JP, Klossek JM, Larenas-Linnemann D, Lipworth B, Malo JL, Marshall GD, Naspitz C, Nekam K, Niggemann B, Nizankowska-Mogilnicka E, Okamoto Y, Orru MP, Potter P, Price D, Stoloff SW, Vandenplas O, Viegi G, Williams D; World Health Organization; GA(2)LEN; AllerGen. Allergic Rhinitis and its Impact on Asthma (ARIA) 2008 update (in collaboration with the World Health Organization, GA(2)LEN and AllerGen). Allergy. 2008 Apr;63 Suppl 86:8-160. doi: 10.1111/j.1398-9995.2007.01620.x. No abstract available. PMID 18331513
- [Result] Alobid I, Anton E, Armengot M, Chao J, Colas C, del Cuvillo A, Davila I, Dordal MT, Escobar C, Fernandez-Parra B, Gras-Cabrerizo JR, Ibanez MD, Lluch M, Mateu V, Montoro J, Gili JR, Mullol J, Navarro AM, Pumarola F, Rondon C, Sanchez-Hernandez MC, Sarandeses A, Soler R, Valero AL; Rhinoconjunctivitis Committee; Spanish Society of Allergy and Clinical Immunology; Rhinology and Allergy Commission; Spanish Society of Otorhinolaryngology. SEAIC-SEORL. Consensus Document on Nasal Polyposis. POLINA Project. J Investig Allergol Clin Immunol. 2011;21 Suppl 1:1-58. No abstract available. PMID 21714471
- [Result] Fokkens WJ, Lund VJ, Mullol J, Bachert C, Alobid I, Baroody F, Cohen N, Cervin A, Douglas R, Gevaert P, Georgalas C, Goossens H, Harvey R, Hellings P, Hopkins C, Jones N, Joos G, Kalogjera L, Kern B, Kowalski M, Price D, Riechelmann H, Schlosser R, Senior B, Thomas M, Toskala E, Voegels R, Wang de Y, Wormald PJ. EPOS 2012: European position paper on rhinosinusitis and nasal polyps 2012. A summary for otorhinolaryngologists. Rhinology. 2012 Mar;50(1):1-12. doi: 10.4193/Rhino12.000. PMID 22469599
- [Result] Chung KF, Wenzel SE, Brozek JL, Bush A, Castro M, Sterk PJ, Adcock IM, Bateman ED, Bel EH, Bleecker ER, Boulet LP, Brightling C, Chanez P, Dahlen SE, Djukanovic R, Frey U, Gaga M, Gibson P, Hamid Q, Jajour NN, Mauad T, Sorkness RL, Teague WG. International ERS/ATS guidelines on definition, evaluation and treatment of severe asthma. Eur Respir J. 2014 Feb;43(2):343-73. doi: 10.1183/09031936.00202013. Epub 2013 Dec 12. PMID 24337046
- [Result] Braunstahl GJ, Fokkens W. Nasal involvement in allergic asthma. Allergy. 2003 Dec;58(12):1235-43. doi: 10.1046/j.0105-4538.2003.00354.x. PMID 14616096
- [Result] Vashishta R, Soler ZM, Nguyen SA, Schlosser RJ. A systematic review and meta-analysis of asthma outcomes following endoscopic sinus surgery for chronic rhinosinusitis. Int Forum Allergy Rhinol. 2013 Oct;3(10):788-94. doi: 10.1002/alr.21182. Epub 2013 Jul 1. PMID 23818462
- [Result] Lildholdt T, Rundcrantz H, Lindqvist N. Efficacy of topical corticosteroid powder for nasal polyps: a double-blind, placebo-controlled study of budesonide. Clin Otolaryngol Allied Sci. 1995 Feb;20(1):26-30. doi: 10.1111/j.1365-2273.1995.tb00007.x. PMID 7788929
- [Result] American Thoracic Society; European Respiratory Society. ATS/ERS recommendations for standardized procedures for the online and offline measurement of exhaled lower respiratory nitric oxide and nasal nitric oxide, 2005. Am J Respir Crit Care Med. 2005 Apr 15;171(8):912-30. doi: 10.1164/rccm.200406-710ST. No abstract available. PMID 15817806
- See also: Guía Española para el Manejo del Asma (GEMA) 4.0 — http://www.gemasma.com